CLINICAL TRIAL: NCT07401836
Title: Can a Standardized Sleep Bundle Reduce Sleep Disruption After Cardiac Surgery: A Pilot Randomized Controlled Trial
Brief Title: Standardized Sleep Bundle for Cardiac Surgery Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Horizon Health Network (Other)
Collaborators: New Brunswick Heart Centre (Other)
Responsible Party: Principal Investigator, Caroline.Fitzpatrick, Principle Investigator, Horizon Health Network
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 102398
Record Dates: First submitted 2026-01-19; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Sleep
Keywords: cardiovascular surgery; sleep

STUDY DESIGN:
Intervention Model Description: Prospective pilot randomized controlled study with a parallel group design comparing a sleep bundle intervention to usual postoperative care, with feasibility as the primary outcome.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sleep Bundle Group (Experimental): Participants in this group will receive a standardized sleep management protocol combining non-pharmacological interventions and stepwise pharmacotherapy.
  Interventions: Other: Standardized Sleep Protocol
- Usual Post Operative Care (Active Comparator): Participants randomized to the control group will receive usual postoperative care.
  Interventions: Other: Usual Post Operative Care

INTERVENTIONS:
Other: Standardized Sleep Protocol — Non-Pharmacological Sleep Aids
  * All participants will be encouraged to wear a sleep mask and ear plugs nightly. In addition, a noise machine will be provided each night, the content and volume of which will be decided by the patient.
  * Stepwise Pharmacotherapy Approach
  Step 1: Melatonin
  - Melatonin 6 mg orally at bedtime will be initiated for all participants in the sleep bundle group.
  Step 2: Adjunctive Therapy (Trazodone)
  * If the participants daily RCSQ score is below 63.4 or the participant reports inadequate sleep despite melatonin, trazodone will be scheduled orally at bedtime.
  * Trazodone will start at 25 mg and may be increased in 25 mg increments up to 100 mg orally at bedtime, based on participant response and tolerability.
  Step 3: Escalation for Delirium (Quetiapine)
  * If the participant has documented postoperative delirium, quetiapine 12.5 mg immediate release oral tablet will be scheduled at bedtime.
  * Dose may be increased in 12.5 mg increments up to 100 mg as cli
  Arms: Sleep Bundle Group
Other: Usual Post Operative Care — Standard postoperative care without the structured sleep bundle. This includes routine clinical management of sleep without non-pharmacological interventions or protocolized pharmacological sleep aid. Any sleep medications administered will be at the discretion of the care team, without a standardized approach, reflecting standard practice.
  Arms: Usual Post Operative Care

SUMMARY:
The goal of this clinical trial is to evaluate the feasibility of using a standardized sleep bundle in adults undergoing cardiac surgery. The main questions it aims to answer are:

1. Can eligible participants be recruited and retained in the study?
2. Can participants follow the study procedures, including using sleep aids and completing daily assessments?
3. Can sleep and other clinical data be reliably collected during the hospital stay? Researchers will compare participants who receive the sleep bundle to participants who receive usual postoperative care.

Participants will:

* Use non-drug sleep aids, including a sleep mask, ear plugs, and a noise machine (sleep bundle group only).
* Take sleep medications if needed, following a stepwise protocol (sleep bundle group only).
* Complete daily sleep assessments using the Richards-Campbell Sleep Questionnaire.
* Wear a Fitbit device at night to track sleep.
* Follow usual postoperative care routines (control group)

The study will also collect and describe data on sleep duration, nighttime awakenings, subjective sleep quality, incidence of postoperative delirium, and hospital length of stay to inform the design of a future larger trial.

DETAILED DESCRIPTION:
This study is a pilot randomized controlled trial designed to evaluate the feasibility and effects of a standardized sleep bundle on sleep quality in patients undergoing cardiac surgery. Adult patients scheduled for non-emergent cardiac surgery at the Saint John Regional Hospital will be screened for eligibility and enrolled after providing informed consent. Participants will be randomized to either usual postoperative care or the sleep bundle group.

The sleep bundle includes non-pharmacological interventions (sleep mask, ear plugs, nightly noise machine) and a stepwise pharmacological approach (melatonin, with trazodone or quetiapine added as needed). Sleep outcomes will be measured objectively using the Fitbit Inspire 3 device and subjectively using the Richards-Campbell Sleep Questionnaire (RCSQ). Feasibility will be assessed based on recruitment, retention, and adherence to the study protocol. Secondary outcomes include total sleep duration, nighttime awakenings, subjective sleep quality, incidence of postoperative delirium, and hospital length of stay.

All study procedures and daily assessments will be conducted by trained research personnel, with data analysis performed by a team member blinded to group allocation. This pilot study will inform the design of a future larger-scale trial.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients over 19 years old, undergoing non-emergent cardiac surgery with cardiopulmonary bypass at the Saint John Regional Hospital (SJRH).

Exclusion Criteria:

* Emergent surgery.
* Severe renal or hepatic impairment (creatinine clearance <30 mL/min, CKD stage ≥4, cirrhosis, ALT ≥ 3× ULN).
* Sleep apnea.
* Restless leg syndrome.
* Insomnia with chronic use of pharmacological sleep aids prior to admission (trazodone, benzodiazepines, zopiclone, mirtazapine, quetiapine, tricyclic antidepressants [nortriptyline, amitriptyline, doxepin]).
* Prior use of a monoamine oxidase inhibitor in the past 14 days.
* QTc > 500ms / history of prolonged QT, Torsade de points or ventricular tachycardia.
* History of dementia, alcohol, or opioid use disorder.
* Documented or previous intolerance to melatonin, trazodone, or quetiapine. Unable to provide informed consent.

Run-in Period Exclusions:

After enrolment and before randomization, participants will be monitored for specific postoperative criteria. Those meeting any of the following criteria will be withdrawn prior to randomization.

* Radial artery harvest required (unable to place Fitbit device on the wrist contralateral to the arterial monitoring line).
* Prolonged intubation or sedation (> 48 hours) post-surgery.
* Major intra- or early postoperative complications (stroke, TIA, major bleeding, need for mechanical/circulatory support, reoperation, open chest, pulmonary embolism, acute renal failure requiring dialysis or other major surgical complications that would inhibit ability to participate).

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-04-17 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Recruitment Rate | From first participant enrollment until last participant enrolled (approximately 8 weeks)
  Proportion of eligible patients who consent to participate in the study. Recruitment success is defined as greater than 50% of eligible patients enrolled. Reported as a percentage.
Retention Rate | From enrollment until hospital discharge for each participant ( approximately 5 days)
  Proportion of participants who complete the study. Retention success is defined as greater than 80% of participants completing the study. Reported as a percentage.
Protocol Adherence | Daily from Day 1 of enrollment through hospital discharge (approximately 5 days)
  Proportion of daily study assessments completed by participants. Reported as a percentage of completed assessments out of total expected assessments.
Fitbit Adherence | Each night from Day 1 of enrollment through hospital discharge (approximately 5 days)
  Number of nights the Fitbit is worn ( minimum 3 scheduled nights). Reported as count and percentage of participants meeting adherence criteria.
Time to Reach Target Sample Size | From first participant enrolment to enrolment of the 20th participant ( approximately 8 weeks)
  Number of days required to enroll the target sample size of 20 participants. Reported in days.

SECONDARY OUTCOMES:
Total Sleep Duration | Nightly from postoperative day 1 through postoperative day 5 or hospital discharge, whichever occurs first.
  Objective sleep duration will be measured using the Fitbit Inspire 3 device, worn on the wrist contralateral to the radial arterial line. The device records total sleep time nightly between 9:00 PM and 9:00 AM. Data will be summarized using daily means, standard deviations, medians, and interquartile ranges.
Nighttime Awakenings | Nightly from postoperative day 1 through postoperative day 5 or until hospital discharge, whichever occurs first
  Objective nighttime awakenings will be measured using the Fitbit Inspire 3 device, recorded nightly between 9:00 PM and 9:00 AM. Daily counts of awakenings will be summarized using means, standard deviations, medians, and interquartile ranges.
Subjective Sleep Quality | Each morning from postoperative day 1 through postoperative day 5 or until hospital discharge, whichever occurs first
  Subjective sleep quality will be assessed each morning using the Richards-Campbell Sleep Questionnaire (RCSQ), a validated 0-100 mm visual analog scale evaluating sleep depth, latency, awakenings, efficiency, and overall quality. Scores will be averaged across the five domains. Daily scores will be summarized using descriptive statistics.
Incidence of Postoperative Delirium | Daily from postoperative day 1 through postoperative day 5 or until hospital discharge, whichever occurs first.
  Incidence of delirium will be recorded based on daily assessments documented by the care team in patient charts. Counts and percentages of participants experiencing delirium will be reported.
Hospital Length of Stay | From day of surgery (postoperative day 0) through postoperative day 5 or until hospital discharge, whichever occurs first
  Length of stay will be recorded in days from the date of surgery to the date of discharge, as documented in the patient's medical record. Data will be summarized using descriptive statistics.

CONTACTS AND LOCATIONS:
Overall Officials: Caroline E Fitzpatrick, Principal Investigator — Horizon Health Network
Locations (1):
- Saint John Regional Hospital, Saint John, New Brunswick, Canada

IPD SHARING:
Plan to Share IPD: Undecided
The decision to share individual participant data has not yet been determined. Plans for data sharing will be considered once the feasibility and outcomes of the pilot study are evaluated.

REFERENCES:
- [Background] Elliott R, Axelin A, Richards KC, Vahlberg T, Ritmala-Castren M. Sensitivity and specificity of proposed Richards-Campbell Sleep Questionnaire cut-off scores for good quality sleep during an ICU stay. J Clin Nurs. 2023 Jun;32(11-12):2700-2708. doi: 10.1111/jocn.16348. Epub 2022 May 15. PMID 35570380
- [Background] Haghayegh S, Khoshnevis S, Smolensky MH, Diller KR, Castriotta RJ. Accuracy of Wristband Fitbit Models in Assessing Sleep: Systematic Review and Meta-Analysis. J Med Internet Res. 2019 Nov 28;21(11):e16273. doi: 10.2196/16273. PMID 31778122
- [Background] Soh PQP, Wong WHT, Roy T, Tam WWS. Effectiveness of non-pharmacological interventions in improving sleep quality after cardiac surgery: A systematic review and meta-analysis. J Clin Nurs. 2024 Jun;33(6):2084-2098. doi: 10.1111/jocn.17115. Epub 2024 Mar 13. PMID 38477050
- [Background] Mahran GS, Leach MJ, Abbas MS, Abbas AM, Ghoneim AM. Effect of Eye Masks on Pain and Sleep Quality in Patients Undergoing Cardiac Surgery: A Randomized Controlled Trial. Crit Care Nurse. 2020 Feb 1;40(1):27-35. doi: 10.4037/ccn2020709. PMID 32006033
- [Background] Liao WC, Huang CY, Huang TY, Hwang SL. A systematic review of sleep patterns and factors that disturb sleep after heart surgery. J Nurs Res. 2011 Dec;19(4):275-88. doi: 10.1097/JNR.0b013e318236cf68. PMID 22089653
- [Background] Simeone S, Pucciarelli G, Perrone M, Teresa R, Gargiulo G, Guillari A, Castellano G, Tommaso LD, Niola M, Iannelli G. Delirium in ICU patients following cardiac surgery: An observational study. J Clin Nurs. 2018 May;27(9-10):1994-2002. doi: 10.1111/jocn.14324. Epub 2018 Apr 25. PMID 29493837
- [Background] Zhang WY, Wu WL, Gu JJ, Sun Y, Ye XF, Qiu WJ, Su CQ, Zhang SQ, Ye WQ. Risk factors for postoperative delirium in patients after coronary artery bypass grafting: A prospective cohort study. J Crit Care. 2015 Jun;30(3):606-12. doi: 10.1016/j.jcrc.2015.02.003. Epub 2015 Feb 7. PMID 25708120
- [Background] Caruana N, McKinley S, Elliott R, Gholizadeh L. Sleep Quality During and After Cardiothoracic Intensive Care and Psychological Health During Recovery. J Cardiovasc Nurs. 2018 Jul/Aug;33(4):E40-E49. doi: 10.1097/JCN.0000000000000499. PMID 29771744